CLINICAL TRIAL: NCT06608199
Title: A Multi-center, Randomized, Blinded, Active-controlled, Phase 3 Clinical Study to Evaluate the Immunogenicity and Safety of 13-valent Pneumococcal Polysaccharide Conjugate Vaccine Co-administered with Hexavalent Vaccine At 2, 4 and 12-15 Months of Age to Healthy Infants in Indonesia
Brief Title: A Phase 3 Study to Evaluate the Immunogenicity and Safety of Minhai's PCV13-DT/TT Vaccine As Compared to Pfizer's PCV13 Vaccine
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Beijing Minhai Biotechnology Co., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: S20210036-5
Record Dates: First submitted 2024-09-19; First posted 2024-09-23 (Actual); Last update posted 2025-03-24 (Actual); Status verified 2025-03

CONDITIONS: Pneumococcal Vaccines; Pneumococcal Infections
Keywords: PCV13; Hexavalent Vaccine; Prevenar 13; Co-administration
MeSH Terms: conditions — Pneumococcal Infections

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- PCV13-DT/TT(Pneuminvac) (Experimental): 250 infants will be administered with Minhai's PCV13-DT/TT(Pneuminvac)
  Interventions: Biological: pneumococcal disease prevention
- PCV13(Prenenar13) (Active Comparator): 250 infants will be administered with Prenenar13
  Interventions: Biological: pneumococcal disease prevention

INTERVENTIONS:
Biological: pneumococcal disease prevention — 2P+1 programme of PCV13

SUMMARY:
The goal of this clinical trial is to evaluate the immunogenicity and safety of Minhai's 13-valent Pneumococcal Polysaccharide Conjugate Vaccine (PCV13-DT/TT) as compared to Pfizer's 13-valent Pneumococcal Conjugate Vaccine (PCV13) when co-administered with Hexavalent Vaccines at 2,4, and 12-15 months of age, to healthy infants in Indonesia. This study aims to demonstrate the non-inferiority of the serotype-specific immune responses elicited by the novel PCV13-DT/TT (Pneuminvac) as compared to PCV13(Prevenar 13) one month after the booster dose, and evaluate the safety of PCV13 co-administrated with Hexavalent Vaccine(Hexaxim).

DETAILED DESCRIPTION:
A total of approximately 500 infants 6-8 weeks of age (WOA) will be enrolled and randomized in 1:1 ratio into the study group and control group, with 250 participants in each group.The study group will receive study PCV13 vaccine and control group will receive Prevenar13® vaccine at 2, 4 and 12-15 months of age (MOA, as early as 6 weeks of age as per WHO recommendations for administration of PCV to infants). Hexavalent vaccine will be injected at 2, 3 and 4 months of age.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy infants based on medical history and clinical assessment.
2. Infants age of 6-8 weeks at enrolment. Infants will be eligible since the day they reach 6 weeks of age and until 8 weeks of age included.
3. *Body weight at enrollment ≥3.0 kg (If the subject does not meet the criteria, the visit may be rescheduled when the criteria is met.).
4. *On the day of vaccination and within 3 days prior to 1st dose of vaccination, axillary temperatures <37.5°C/99.1°F (If the subject does not meet the criteria, the visit may be rescheduled when the criteria is met.).
5. Infant's parent(s) or legal guardian must be able and willing to provide voluntary written/thumb-printed informed consent for the infant to participate in the study.
6. Infant's parent(s) or legal guardian must be willing and able to comply with all scheduled visits, vaccination plan, laboratory tests, lifestyle considerations, and other study procedures.
7. The infant's mother must provide related medical certificate(s) for the negative results for HIV, HBV and syphilis infection within 1 year prior to screening.
8. Infant's parent(s) or legal guardian must have a readily identifiable place of residence in the study area, be available for the duration of trial participation, and have a means of telephone contact.

Note: For items with an asterisk (*), If the subject does not meet the criteria, the visit may be rescheduled when the criteria is met.

Exclusion Criteria:

1. Use of any investigational product other than that used in the study prior to randomization or planned use of such a product during the period of study participation.
2. History of S. pneumoniae infection as confirmed by laboratory testing if available.
3. The infant who are children in care, preterm and low-birth-weight (Preterm infants have a gestational age below 37 weeks at birth and low-birth-weight infants have a birth weight below 2.5 kg).
4. History of allergic disease or history of a serious reaction to any prior vaccination or known hypersensitivity to any component of the investigational vaccine. And/or all components of the hexavalent vaccine.
5. History of anaphylactic shock.
6. Any abnormal vital sign as judged by the investigator.
7. *Participant experiences acute diseases or acute exacerbation of chronic diseases or uses antipyretic, analgesic and anti-allergic drugs (such as paracetamol, ibuprofen, aspirin, loratadine, cetirizine, etc.) within 3 days before vaccination.
8. *History of administration of attenuated vaccines within 14 days (<14 days) and inactivated vaccines within 7 days (<7 days) prior to the 1st dose of investigational vaccine (If the participant[s] does not meet the criteria, the visit may be rescheduled when the criteria are met).
9. Previous vaccination against diphtheria, tetanus, pertussis, polio, hepatitis B, Haemophilus influenzae type b, Neisseria meningitidis and/or Streptococcus pneumoniae with the exception of vaccines where the first dose can be given before 2 months of life according to the national recommendations.
10. History of or intercurrent diphtheria, tetanus, pertussis, hepatitis B, polio, Haemophilus influenzae type b disease, Neisseria meningitidis.
11. Individuals who receive treatment with radiotherapy or immunosuppressive therapy, including cytotoxic agents or systemic corticosteroids (if systemic corticosteroids are administered for ≥14 days at a dose of ≥10 mg/day of prednisone or equivalent), e.g., for cancer or an autoimmune disease, or planned receipt throughout the study. Inhaled/nebulized, intra-articular, epidural, or topical (skin or eyes) corticosteroids within indicated dosage are permitted.
12. *Administration of immunoglobulins and/or any blood products or anticipation of such administration within 28 days before vaccination and during the study period.
13. History of known disturbance of coagulation or blood disorder that could cause anemia or excess bleeding (e.g., thalassemia, coagulation factors deficiency, severe anemia at birth).
14. History of suspected primary immunodeficiency.
15. History of meningitis, seizures or any neurological disorder.
16. A family history of congenital or hereditary immunodeficiency.
17. The infant is a direct descendant (child or grandchild) of any person employed by the Sponsor, the CRO, the investigator, study site personnel.
18. Any medical or social condition that in the opinion of the investigator may compromise the well-being of the study participant, interfere with the study objectives, pose a risk to the study participant, or prevent the study participant from completing the study follow-up.

Note: For items with an asterisk (*), if the participant meets these exclusion criteria, the visit may be rescheduled for a time when these criteria are not met.

Ages: 6 Weeks to 8 Weeks | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 500 (Estimated)
Dates: Start 2024-11-01 (Actual); Primary Completion 2025-06-01 (Estimated); Study Completion 2026-10-01 (Estimated)

PRIMARY OUTCOMES:
Immugenocity | 1. Percentage of participants with serotype-specific IgG concentrations ≥ 0.35 μg/mL, measured 30 days after the booster dose of the investigational vaccine. 2. GMC ratio of serotype-specific IgG responses 30 days after the booster dose of the investigat
  1. To evaluate the serotype-specific IgG responses 30 days after booster dose of the investigational vaccine.

SECONDARY OUTCOMES:
Safety | 1.Incidence, severity and duration of each solicited (local and systemic) AE within 7 days after each dose of the investigational vaccine in all participants.
  1.To assess the solicited AEs (local and systemic) occurring 0-7 days after each dose of the investigational vaccine.
Safety | 2. Incidence, severity, and causality of unsolicited AEs within 30 days after each dose of the investigational vaccine in all participants.
  2. To assess the unsolicited AEs occurring 0-30 days after each dose of the investigational vaccine.
Safety | 3. Incidence, severity, and causality of SAEs from 1st dose to 6 months after booster dose of the investigational vaccine.
  3. To assess SAE from 1st dose to 6 months after booster dose of the investigational vaccine.
Immugenocity | 1. Percentage of participants with serotype-specific IgG concentrations ≥ 0.35 μg/mL, measured 30 days after 2nd dose of the investigational vaccine. 2. GMC of serotype-specific IgG responses 30 days after 2nd dose of the investigational vaccine. 3. Pe
  1. To evaluate the serotype-specific IgG responses 30 days after 2nd dose of the investigational vaccine.
  2. To evaluate the serotype-specific Opsonophagocytic Activicity (OPA) 30 days after the 2nd dose, before the booster dose, and 30 days after the booster dose of the investigational vaccine in OPA subgroup.
  3. To evaluate the immune responses induced by hexavalent vaccine 30 days after the 2nd dose of the investigational vaccine in different subsets.

CONTACTS AND LOCATIONS:
Locations (3):
- Indonesia (3):
  - Faculty of Medicine Udayana University, Denpasar, Bali
  - Universitas Padjadjaran Bandung, Bandung, Bandung
  - Faculty of Medicine, padjadjaran University, Bandung, Bandung

IPD SHARING:
Plan to Share IPD: No